CLINICAL TRIAL: NCT03556189
Title: Effect of Atrioventricular Optimization on Left Ventricular Function With Dual Chamber Pacemaker; Prospective Randomized Trial
Brief Title: Atrioventricular Optimization for Dual Chamber Pacemaker
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yong Seog Oh (Other)
Responsible Party: Sponsor-Investigator, Yong Seog Oh, professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AV delay
Record Dates: First submitted 2017-04-24; First posted 2018-06-14 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: AV Block
MeSH Terms: conditions — Atrioventricular Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): case management consists adjusting AV delay of pacemaker to achieve best cardiac output measured by trans-thoracic echocardiogram
  Interventions: Device: Case management
- Control: Usual care (No Intervention): Usual care is provided with routine pacemaker interrogation.

INTERVENTIONS:
Device: Case management — Case management consists adjusting AV delay of pacemaker to achieve best cardiac output measured by trans-thoracic echocardiogram
  Arms: Experimental

SUMMARY:
This study aims to examine the effect of atrioventricular synchrony in AV block patients who received permanent pacemaker. By achieving physiologic ventricular diastolic filling, adjustment of atrioventricular delay of pacemaker might affect the long term outcome of left ventricular function and remodelling. The investigators designed to randomize AV block patients who already have or anticipated to receive pacemaker, into two groups. Patients in intervention group undergo reprogramming AV delay of pacemaker to the best value to increase cardiac output measured by transthoracic echocardiogram and the patients in control group undergo routinely scheduled pacemaker programming. The primary endpoint is improvement of LV systolic function and the secondary endpoint is change in left ventricular volume, cardiac output, BNP, 6-minute walk capacity and NYHA class after one year.

DETAILED DESCRIPTION:
It is well-known that persistent right ventricular apical pacing induces left ventricular dysfunction. The most important risk factor is the ratio of ventricular pacing so the effort to reduce pacing ratio is needed. However, almost 100% ventricular pacing is inevitable in complete atrio-ventricular block patients with implanted pacemaker. Traditionally the ventricular lead of the pacemaker is positioned in right ventricular apex and previous literatures reported that such right ventricular apical pacing impedes physiological ventricular contraction and induces left ventricular contractile dysfunction in long-term. The alternative positions of ventricular lead are right ventricular outflow tract and ventricular septum but the benefits are not yet clearly prooved. Additionally, adjusting atrio-ventricular delay is reportedto affect cardiac output by altering diastolic filling. The investigators aimed to analyze the effect of AV dealy in long-term left ventricular contractile function.

Patients over 19 years old who received or anticipated to receive permanent pacemaker due to AV block are randomized to 1:1 ratio into two groups. Patients in intervention group undergo reprogramming AV delay of pacemaker to the best value to increase cardiac output measured by transthoracic echocardiogram and the patients in control group undergo routinely scheduled pacemaker programming. Patients with underlying LV systolic dysfunction or significant valvular heart disease are excluded. Six-minute walk test, BNP, transthoracic echocardiogram, NYHA class are examined at baseline and after one year.

ELIGIBILITY:
Inclusion Criteria:

* Received or scheduled to receive permanent pacemaker due to AV block

Exclusion Criteria:

* Left ventricular ejection fraction <50% or Left ventricular end-diastolic diameter>60mm Significant valvular disease (≥mild)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | one year after randomization

SECONDARY OUTCOMES:
Left ventricular end-diastolic diameter | one year after randomization
Left ventricular end-systolic diameter | one year after randomization
cardiac output | one year after randomization
BNP | one year after randomization
6-minute walking test | one year after randomization
NYHA class | one year after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Seog Oh, MD,PhD, Principal Investigator — The Catholic University of Korea
Locations (1):
- Seoul St Mary's Hospital, Seoul, Seo Ch-gu, South Korea